CLINICAL TRIAL: NCT02003963
Title: Klub Kinect: Social Exergaming for Healthy Weight in Adolescent Girls
Brief Title: Social Exergaming for Healthy Weight in Adolescent Girls
Acronym: Klub Kinect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 2013-046
Record Dates: First submitted 2013-11-26; First posted 2013-12-06 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Obesity and Physical Inactivity in Adolescents
Keywords: Physical Activity; Sedentary Behavior; Video Games; Exergames
MeSH Terms: conditions — Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame Intervention (Experimental): Participants randomly assigned to the exergame condition will participate in the intervention condition of "Klub Kinect." Klub Kinect is a 12-week intervention occurring for 90-minute sessions, 3 times per week. During each 90-minute intervention session, adolescents will engage in 60-minute bouts of aerobic gaming. Adolescents attending an exergaming session will attend concurrently.
  Interventions: Behavioral: Klub Kinect
- Control (Self-Directed Care) (No Intervention): The control condition will receive no contact or intervention other than telephone reminders of their final clinic visit.

INTERVENTIONS:
Behavioral: Klub Kinect — Dance Central and Just Dance are a series of rhythm games developed by Harmonix Music Systems exclusively for the Xbox 360 Kinect. The Dance Central suite of games (Dance Central 1, 2, and 3) and Just Dance will be played on the Xbox 360+ Kinect gaming console, which employs whole body movement using an infrared sensor that tracks body movements such that an external controller device is not required. The player performs dance moves demonstrated by on-screen characters and set to popular music, with a choice of over 650 dance moves, 90 dance routines, and over 300 songs.
  The exergaming condition will wear a pedometer to record total steps during game play, and they will participate in private weigh-ins at each session to track body weight over the 12-week intervention.
  Arms: Exergame Intervention

SUMMARY:
The purpose is to evaluate the feasibility of a 12-week exergaming dance program for adolescent girls. This study combines dancing, video games, and a full body work-out to test if video games can increase physical activity and promote healthy weight in adolescent girls. We hypothesize that girls who play the dance exergames, versus those in the control group, will lose weight, decrease body fat and visceral fat, improve cardiovascular health, increase physical activity, and improve psychosocial health including self-confidence and quality of life.

DETAILED DESCRIPTION:
Klub Kinect will last about 14 weeks for each participant. The program begins with a 3.5 hour clinic visit, the intervention lasts for 12 weeks, and the participant comes in for a final 3.5 hour clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18 years old
* Female
* Postmenarchal
* BMI percentile equal to or greater than 85th on the U.S. Centers for Disease Control and Prevention growth chart
* Speak, understand, read, and write English
* Willing to accept randomization

Exclusion Criteria:

* Pregnant
* Hospitalization for mental illness within the past 5 years.
* Since the focus herein is on ambulatory activities, participants who use wheelchairs or other impairments that prevent normal ambulation will be excluded
* Indication of cardiac abnormality on an electrocardiogram that requires referral to a cardiologist
* Previous history of, or clinical symptoms or signs of, cardiovascular disease, stroke or transient ischemic attacks, chest pain, unusual dyspnea during physical activity/exercise, severe ankle edema, or intermittent claudication.
* Previous history of musculoskeletal injuries or problems causing severe pain during physical activity or exercise which interferes with daily activities.
* Participant has a pacemaker or other implanted medical device (including metal joint replacements).
* Participant is unable to complete all baseline testing (one session) within 1 month prior to the beginning of the intervention
* Medical problems, including epileptic seizures, that prevent video game play
* Family history of epileptic seizures
* Unable to make the commitment of coming to Pennington Biomedical Research Center for 3 weekly gaming sessions for 12 weeks

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Staiano AE, Marker AM, Beyl RA, Hsia DS, Katzmarzyk PT, Newton RL. A randomized controlled trial of dance exergaming for exercise training in overweight and obese adolescent girls. Pediatr Obes. 2017 Apr;12(2):120-128. doi: 10.1111/ijpo.12117. Epub 2016 Feb 26. PMID 26918815
- [Result] Staiano AE, Beyl RA, Hsia DS, Katzmarzyk PT, Newton RL Jr. Twelve weeks of dance exergaming in overweight and obese adolescent girls: Transfer effects on physical activity, screen time, and self-efficacy. J Sport Health Sci. 2017 Mar;6(1):4-10. doi: 10.1016/j.jshs.2016.11.005. Epub 2016 Nov 23. PMID 28491483
- [Result] Staiano AE, Beyl RA, Hsia DS, Katzmarzyk PT, Newton RL Jr. A 12-week randomized controlled pilot study of dance exergaming in a group: Influence on psychosocial factors in adolescent girls. Cyberpsychology (Brno). 2018;12(2):3. doi: 10.5817/CP2018-2-3. PMID 31367239
- See also: Participant registration — http://www.pbrc.edu/klubkinect

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overweight and obese adolescent girls were recruited for study participation. Participants were screened and enrolled at Pennington Biomedical Research Center. 200 adolescents expressed interest in the study.
Groups:
- Exergame Intervention: Participants randomly assigned to the exergame condition will participate in the intervention condition of "Klub Kinect." Klub Kinect is a 12-week intervention occurring for 90-minute sessions, 3 times per week. During each 90-minute intervention session, adolescents will engage in 60-minute bouts of aerobic gaming. Adolescents attending an exergaming session will attend concurrently.
  Klub Kinect: Dance Central and Just Dance are a series of rhythm games developed by Harmonix Music Systems exclusively for the Xbox 360 Kinect. The Dance Central suite of games (Dance Central 1, 2, and 3) and Just Dance will be played on the Xbox 360+ Kinect gaming console, which employs whole body movement using an infrared sensor that tracks body movements such that an external controller device is not required. The player performs dance moves demonstrated by on-screen characters and set to popular music, with a choice of over 650 dance moves, 90 dance routines, and over 300 songs.
Period: Overall Study
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Started | 22 | 19
Completed | 20 (2 participants dropped out: 1 due to lack of interest and 1 due to a mental health hospitalization.) | 18 (1 participant was removed from analysis for completing final visit outside of visit window.)
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exergame Intervention | Control (Self-Directed Care) | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.2) | 16.1 (1.4) | 15.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41
Weight [Mean (Standard Deviation); unit: kilograms] | 97.2 (27.3) | 101.1 (26.1) | 99.15 (26.7)
Height [Mean (Standard Deviation); unit: centimeters] | 160.4 (5.9) | 164.9 (5.8) | 162.65 (5.9)
BMI (z-score) [Mean (Standard Deviation); unit: Z-score] | 2.1 (0.5) | 2.1 (0.5) | 2.1 (0.5)
BMI (percentile) [Mean (Standard Deviation); unit: Percentile] | 97.4 (2.9) | 97.1 (3.3) | 97.3 (3.1)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] | 107.3 (22.0) | 107.7 (21.1) | 107.5 (21.6)
DXA Total body fat [Mean (Standard Deviation); unit: kilograms] | 47.0 (19.7) | 48.0 (17.0) | 47.5 (18.35)
DXA Total body fat percent [Mean (Standard Deviation); unit: percentile] | 48.3 (19.7) | 48.2 (6.3) | 48.25 (13)
DXA leg fat [Mean (Standard Deviation); unit: kilograms] | 16.2 (5.6) | 16.2 (4.7) | 16.2 (5.2)
DXA Leg fat percentage [Mean (Standard Deviation); unit: percentile] | 48.3 (5.6) | 48.0 (5.2) | 48.2 (5.4)
DXA Gynoid Fat [Mean (Standard Deviation); unit: kilograms] | 7.6 (2.5) | 8.1 (2.2) | 7.9 (4.7)
DXA Gynoid Fat Percentage [Mean (Standard Deviation); unit: Percentile] | 49.8 (6.5) | 50.1 (4.9) | 50 (5.7)
DXA Android Fat [Mean (Standard Deviation); unit: Kilograms] | 4.2 (2.2) | 4.4 (2.3) | 4.3 (2.3)
DXA Android Fat Percentile [Mean (Standard Deviation); unit: Percentile] | 53.8 (10.5) | 54.3 (9.2) | 54.1 (19.7)
DXA Trunk Fat [Mean (Standard Deviation); unit: Kilograms] | 25.1 (13.6) | 26.1 (12.1) | 25.6 (12.9)
DXA Trunk Fat Percentile [Mean (Standard Deviation); unit: Percentile] | 50.6 (9.5) | 50.5 (8.1) | 50.6 (8.8)
DXA Bone Mineral Content (BMC) [Mean (Standard Deviation); unit: Kilograms] | 2.6 (0.3) | 2.7 (0.3) | 2.65 (0.3)
DXA Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: Grams per centimeter squared] | 1.2 (0.1) | 1.2 (0.1) | 1.2 (0.1)
DXA BMD Trunk [Mean (Standard Deviation); unit: Grams per centimeter squared] | 1.1 (0.1) | 1.1 (0.1) | 1.1 (0.1)
DXA BMD Spine [Mean (Standard Deviation); unit: Grams per centimeter squared] | 1.1 (0.1) | 1.2 (0.1) | 1.15 (0.1)
DXA BMD Leg [Mean (Standard Deviation); unit: Grams per centimeter squared] | 1.3 (0.1) | 1.3 (0.1) | 1.3 (0.1)
MRI Visceral Adipose Tissue [Mean (Standard Deviation); unit: Kilograms] — Population: The sample did not include 3 participants who did not undergo the MRI scan due to exceeding weight limits for the MRI machine or having a metal object in the body.
  Kilograms
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 1.0 (0.7) | 1.0 (0.7) | 1.0 (0.7)
MRI Subcutaneous Adipose Tissue [Mean (Standard Deviation); unit: Kilograms] — Population: The sample did not include 3 participants who did not undergo the MRI scan due to exceeding weight limits for the MRI machine or having a metal object in the body.
  Kilograms
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 12.1 (5.6) | 12.3 (5.7) | 12.2 (5.65)
MRI Total Adipose Tissue [Mean (Standard Deviation); unit: Kilograms] — Population: The sample did not include 3 participants who did not undergo the MRI scan due to exceeding weight limits for the MRI machine or having a metal object in the body.
  Kilograms
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 13.1 (5.9) | 13.3 (6.3) | 13.2 (6.1)
Systolic Blood Pressure Percentile [Mean (Standard Deviation); unit: Percentile] | 63.5 (25.2) | 56.6 (30.1) | 60.1 (27.7)
Diastolic Blood Pressure Percentile [Mean (Standard Deviation); unit: Percentile] | 60.9 (22.3) | 66.4 (20.5) | 63.7 (21.4)
Cholesterol [Mean (Standard Deviation); unit: Milligrams per deciliter] | 149.6 (21.6) | 163.1 (27.3) | 156.6 (24.5)
High Density Lipoprotein [Mean (Standard Deviation); unit: Milligrams per deciliter] | 47.4 (7.3) | 52.7 (10.5) | 50.1 (8.9)
Low-density Lipoprotein [Mean (Standard Deviation); unit: Milligrams per deciliter] | 86.4 (19.2) | 94.4 (22.9) | 90.4 (21.1)
Triglycerides [Mean (Standard Deviation); unit: Milligrams per deciliter] | 78.9 (49.4) | 80.0 (42.4) | 79.5 (45.9)
Glucose [Mean (Standard Deviation); unit: Milligrams per deciliter] | 87.6 (6.4) | 91.8 (21.8) | 89.7 (28.2)
Insulin [Mean (Standard Deviation); unit: Micro unit per milliliter] | 24.2 (15.2) | 19.4 (10.4) | 21.8 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Fat
Description: Assessed by dual energy x-ray absorptiometry
Time Frame: Baseline clinic visit (week 0) and final clinic visit (week 13)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Exergame Intervention: Participants randomly assigned to the exergame condition will participate in the intervention condition of "Klub Kinect." Klub Kinect is a 12-week intervention occurring for 90-minute sessions, 3 times per week. During each session, adolescents will engage in 60-minute bouts of aerobic gaming. Adolescents attending an exergaming session will attend concurrently.
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 22 | 19
kg | 1.0 (0.5) | 1.6 (0.5)

2. Primary Outcome: Change in Visceral Adiposity
Description: Assessed by magnetic resonance imaging
Time Frame: Baseline clinic visit (week 0) and final clinic visit (week 13)
Population: Intent to treat. Three participants did not complete baseline or final MRI scan due to exceeding weight limit or metal-containing object in the body, and five participants refused to complete final MRI scan.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 18 | 15
kg | 0.02 (0.03) | 0.04 (0.03)
Statistical Analysis 1: Comparison: Exergame Intervention vs Control (Self-Directed Care); Test type: Superiority; p = 0.05, ANCOVA

3. Primary Outcome: Change in Resting Systolic Blood Pressure Percentile
Description: Resting systolic blood pressure percentile
Time Frame: Baseline clinic visit (week 0) and final clinic visit (week 13)
Measure: Mean (Standard Deviation); unit: %ile
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 20 | 18
%ile | -13.3 (6.3) | -1.8 (6.4)

4. Secondary Outcome: Feasibility (Adherence)
Description: Attendance to exergaming intervention
Time Frame: 3 gaming sessions/week for 12 weeks
Population: Attendance was only assessed for the "Exergame Intervention" participants
Measure: Mean (Full Range); unit: percentage exergaming sessions attended
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 22 | 19
percentage exergaming sessions attended | 79 [28 to 100] | NA [NA to NA] — Attendance was only assessed for the "Exergame Intervention" participants

5. Secondary Outcome: Change in Physical Activity
Description: Actigraph accelerometer (7-day protocol using waking hours) and self-report instrument
Time Frame: Baseline clinic visit (week 0) and final clinic visit (week 13)
Population: Data reported on participants with complete accelerometry data
Measure: Mean (Full Range); unit: change in self-reported days/week of PA
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 19 | 18
change in self-reported days/week of PA | 1.0 [-7 to 7] | -0.3 [-7 to 7]

6. Secondary Outcome: The Friendship Quality Questionnaire to Measure Change in Peer Support From Baseline to Week 13.
Description: The outcome is perceived peer conflict from the Friendship Quality Questionnaire, which is a 21-item self-report survey in which the participant answers questions about his or her best friend related to companionship, conflict, help/aid, security, and closeness, on a 5-point Likert scale. The survey is internally consistent, with α ranging from 0.71 to 0.86, and adequate criterion validity across sub-scales. The peer conflict sub-scale includes four questions and ranges from 4 to 20 points. A higher score indicates higher (worse) levels of peer conflict.
Time Frame: Baseline clinic visit (week 0) and final clinic visit (week 13)
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 22 | 19
change in units on a scale | -0.4 (0.7) | 1.7 (0.7)

7. Secondary Outcome: Change From Baseline in Health-related Quality of Life
Description: Self-report instrument to capture health-related quality of life (KIDSCREEN-10 Index). The scale ranges from 5 to 50, with a higher score indicating a better quality of life.
Time Frame: Baseline clinic visit (week 0) and final clinic visit (week 13)
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 22 | 19
change in units on a scale | -0.1 (1.5) | -1.3 (1.6)

8. Secondary Outcome: Change From Baseline in Self-efficacy Towards Exercise on the Self-Efficacy for Healthy Eating and Physical Activity Measure (SE-HEPA) at Week 13
Description: SE-HEPA is a 13-item self-report survey with items based on a 5-point Likert scale. Possible scores range from 1 (Disagree a Lot) to 5 (Agree a Lot). The items are summed to a total score, and a higher score indicates a higher level of self-efficacy (range: 13 to 65). Results are reported as change scores from baseline.
Time Frame: Baseline clinic visit (Week 0) and final clinic visit (Week 13)
Population: Four participants refused to complete the final assessment.
Measure: Mean (Standard Deviation); unit: change scores on a scale
Groups:
- Exergame Intervention: Klub Kinect is a 12-week intervention occurring for 90-minute sessions, 3 times per week. During each 90-minute intervention session, adolescents will engage in 60-minute bouts of aerobic gaming. Adolescents attending an exergaming session will attend concurrently.
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
Number analyzed (Participants) | 19 | 18
change scores on a scale | 0.37 (1.7) | 0.44 (1.7)

ADVERSE EVENTS:
Time Frame: 8 months (entire duration of the study)
Arm/Group | Exergame Intervention | Control (Self-Directed Care)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No